CLINICAL TRIAL: NCT03406650
Title: Neoadjuvant and Adjuvant Durvalumab in Combination With Neoadjuvant Chemotherapy in Patients With Operable Urothelial Cancer. A Multicenter, Single-arm Phase II Trial
Brief Title: Neoadjuvant and Adjuvant Durvalumab in Combination With Neoadjuvant Chemotherapy in Patients With Operable Urothelial Cancer.
Acronym: SAKK 06/17
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 06/17; 2017-003565-10 (EudraCT Number)
Record Dates: First submitted 2017-12-22; First posted 2018-01-23 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Cancer
Keywords: muscle invasive urothelial cancer; cancer; immunotherapy; durvalumab; MEDI4736; adjuvant; neoadjuvant; radical cystectomy; bladder
MeSH Terms: conditions — Neoplasms | interventions — Neoadjuvant Therapy; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab in combination with standard therapy (Experimental): Combination of standard therapy consisting (4 cycles cisplatin/ gemcitabin followed by surgery) with 4 cycles of neoadjuvant durvalumab and 10 cycles of adjuvant durvalumab
  Interventions: Drug: Neoadjuvant and adjuvant durvalumab

INTERVENTIONS:
Drug: Neoadjuvant and adjuvant durvalumab — Neoadjuvant durvalumab 1500 mg q3w for 4 cycles Adjuvant durvalumab 1500 mg q4w for 10 cycles
  Other Names: MEDI4736

SUMMARY:
The main objective is to demonstrate that the addition of neoadjuvant and adjuvant immunotherapy with durvalumab, to standard neoadjuvant chemotherapy (with cisplatin/gemcitabine) and surgery in urothelial carcinoma could improve event-free survival.

DETAILED DESCRIPTION:
Despite optimal surgical management the prognosis for localized muscle invasive urothelial cancer (MIUC) is unfavorable with 5-year overall survival of around 45%.

According to international guidelines the use of cisplatin-based neoadjuvant chemotherapy is considered standard of care in all patients with localized MIUC with planned curative local treatment.

However, the benefit of neoadjuvant chemotherapy is limited and there is a clear medical need for improvement for this patient population.

Durvalumab has been tested in a phase I/II open-label study including patients with metastatic urothelial cancer (mUC).

The results demonstrated an overall response rate (RR) of 31% in 42 response-evaluable patients. The side effect profile was favorable with most common grade 1/2 AE representing fatigue (13%), diarrhea (10%) and decreased appetite (8%). Three patients (4.9%) had treatment related grade 3 AE's, no grade 4/5 events were noted.

The combination of cisplatin/gemcitabine chemotherapy with modern immune-checkpoint inhibition has been demonstrated to be feasible with demonstration of favorable immunomodulatory effects.

In view of these data it appears a logical step to apply these novel agents in the curative setting of neoadjuvant treatment.

The expected benefit of combining chemotherapy with durvalumab and to continue durvaluamb postoperatively might be twofold:

* to increase the response rate in the pre-operative setting and subsequently to increase the rate of pathologic complete remission (pT0) and to reduce risk of local recurrence
* to evoke durable systemic anti-cancer responses and subsequently to increase disease free- and overall survival and furthermore to induce antitumor immune response.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures
* Histologically proven urothelial cell carcinoma of the bladder, urethra or upper urinary tract (T2, T3, or T4a and ≤ N1 (defined as a solitary lymph node ≤ 2 cm in the greatest dimension), M0) and be considered suitable for curative multimodality treatment including surgery by a multidisciplinary tumor board. Cytological diagnosis is only allowed for upper tract urothelial carcinoma. In these cases tumor has to be documented by urography
* All histological subtypes eligible if urothelial carcinoma predominant (exception: small cell component)
* Age ≥ 18 years
* WHO performance status 0-1
* Bone marrow function: hemoglobin ≥ 90 g/L, neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L
* Hepatic function: bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), AST ≤ 2.5 x ULN and ALT ≤ 2.5 x ULN, alkaline phosphatase ≤ 2.5 x ULN
* Renal function: estimated glomerular filtration rate (eGFR) > 50 mL/min/1.73m², according to CKD-EPI formula
* Cardiac function: Left ventricular Ejection Fraction (LVEF) ≥ 50% as determined by echocardiography (ECHO)
* Women with child-bearing potential are using effective contraception (for details of definition see 9.9), are not pregnant or lactating and agree not to become pregnant during trial treatment and during 90 days thereafter. A negative pregnancy test before inclusion into the trial is required for all women with child-bearing potential
* Men agree not to father a child during trial treatment and during 90 days thereafter
* Body weight > 30kg.

Exclusion Criteria:

* Any pathological evidence of small-cell carcinoma component
* Presence of any distant metastasis
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years before registration, with the exception of adequately treated cervical carcinoma in situ, localized non-melanoma skin cancer or low risk localized prostate cancer (T1-T2a, Gleason <7, PSA <10ng/ml)
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including durvalumab
* Concurrent treatment with prednisone (or equivalent); except for the prophylactic medication before chemotherapy, treatment of acute hypersensitivity reactions or chronic treatment (initiated > 6 months prior to registration) at low dose (≤ 10 mg/day of prednisone or an equivalent corticosteroid)
* Concurrent treatment with other experimental drugs or other anticancer therapy, treatment in a clinical trial within 28 days prior to registration
* Current or prior use of immunosuppressive medication within 28 days prior to registration, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids
* Major surgical procedure within 28 days prior to registration
* Preexisting peripheral neuropathy (> grade 1)
* Uncontrolled diabetes mellitus
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the coordinating investigator
  * Patients with celiac disease controlled by diet alone
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment
* History of allogeneic organ transplant
* Receipt of live attenuated vaccine within 30 days prior to registration. Note: Patients, if enrolled, should not receive live vaccine during trial treatment and up to 30 days after the last dose
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Any concurrent drug contraindicated for blocking the effect of durvalumab; this includes systemic corticosteroids, methotrexate, azathioprine, and tumor necrosis factor (TNF)-α blockers. Any concurrent drug contraindicated for use with the other trial drugs according to the locally approved product information
* Known hypersensitivity to cisplatin, gemcitabine or durvalumab or to any excipient
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
event-free survival (EFS) | 2 years after treatment start
  The primary endpoint of the trial is Event-free survival (EFS) at 2 years after neoadjuvant trial treatment start.
  Event-free survival is defined as the time from treatment start until one of the following events, whichever comes first:
  * Progression during neoadjuvant treatment leading to inoperability
  * Recurrence of locoregional disease after surgery
  * Appearance of metastases at any localization
  * Death Patients not experiencing an event will be censored at the date of the last available assessment before initiation of a subsequent treatment, if any.

SECONDARY OUTCOMES:
Event-free survival (EFS) | at the occurrence of the event or latest 5 years after surgery
  Event-free survival is defined as the time from treatment start until one of the following events, whichever comes first:
  * Progression during neoadjuvant treatment leading to inoperability
  * Recurrence of locoregional disease after surgery
  * Appearance of metastases at any localization
  * Death Patients not experiencing an event will be censored at the date of the last available assessment before initiation of a subsequent treatment, if any.
Recurrence-free survival (RFS) after R0 resection | at recurrence or latest 5 years after surgery
  RFS after R0 resection is defined as the time from surgery until one of the following events, whichever comes first:
  * Recurrence of locoregional disease
  * Appearance of metastases at any localization
  * Death Patients not experiencing an event will be censored at the date of the last available assessment before initiation of a subsequent treatment, if any.
  This endpoint will only be calculated for patients in the R0 resection set.
Overall survival (OS) | at death or latest 5 years after surgery
  Overall survival is defined as the time from treatment start until death from any cause. Patients not experiencing an event will be censored at the last date they were known to be alive.
Quality of resection | after surgery or the latest 20 weeks after registration
  The quality of resection will be assessed in the following way:
  * Complete resection (R0) defined as free resection margins proved microscopically
  * Completeness of the lymphadenectomy and surgery using the photo documentation and histopathology
  * Postoperative complications will be assessed using the Clavien-Dindo classification
Pathological complete response rate (ypT0) | after surgery or the latest 20 weeks after registration
  Pathological complete response (ypT0) is defined as no residual tumor in the surgical specimen. The proportion of patients with ypT0 will be calculated for patients in the resected patients set.
Pathological response rate (PaR) defined by pathological downstaging to ≤ypT1N0M0 | after surgery or the latest 20 weeks after registration
  Pathological response (PaR) is defined as pathological downstaging to ≤ ypT1N0M0. The proportion of patients with PaR will be calculated for patients in the resected patients set.
Pattern of recurrence | after recurrence or latest 5 years after surgery
  Pattern of recurrence is defined as location of first tumor recurrence. Patterns can be locoregional or distant or any combination of these patterns.
  Patients with secondary malignancies or patients with no recurrence will not be taken into consideration for this endpoint.
Treatment feasibility | after treatment end or the latest 73 weeks after registration
  The following feasibility criteria will be assessed:
  * completion of 4 cycles of neoadjuvant chemotherapy
  * completion of 4 cycles of neoadjuvant durvalumab treatment
  * timely admission to and completion of planned surgery
  * timely initiation and completion of 10 cycles of adjuvant durvalumab treatment
Adverse events | within treatment start and 90 days after last trial treatment and resolution of all related AEs thereafter (at the latest 5 years after surgery)
  All AEs will be assessed according to NCI CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cathomas, MD, Study Director — Kantonsspital Graubünden, Chur
Locations (17):
- Germany (2):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Urologische Universitätsklinik Essen, Essen
- Switzerland (15):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - Inselspital, Bern
  - Kantonsspital Graubünden, Chur
  - Spital Thurgau AG, Frauenfeld
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden - Onkozentrum Hirslanden, Zurich
  - OnkoZentrum Zürich, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No